CLINICAL TRIAL: NCT00957060
Title: A Multicenter, Open, Randomized, 24 Weeks Study to Evaluate the Superiority of Glimepiride Over Sitagliptin for the Treatment of naïve Patients With Type 2 Diabetes Mellitus
Brief Title: Superiority of Glimepiride Over Sitagliptin in Naive Type 2 Diabetes Patients
Acronym: SUMER
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Trial Transparency Team, sanofi-aventis
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GLIME_L_04140
Record Dates: First submitted 2009-08-11; First posted 2009-08-12 (Estimated); Last update posted 2010-11-30 (Estimated); Status verified 2010-11

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — glimepiride; Sitagliptin Phosphate

ARMS (2):
- glimepiride (Experimental): The initial dose is 2 mg once a day. At week 2, the dose can be increased to 4 mg once a day according to the titration. At week 4 and 12, the dose can be increased from 2 mg to 4 mg or from 4 mg to 6 mg according to the titration.
  Interventions: Drug: GLIMEPIRIDE (HOE490)
- sitagliptin (Active Comparator): 100 mg once a day. The dose will not be titrated.
  Interventions: Drug: SITAGLIPTIN

INTERVENTIONS:
Drug: GLIMEPIRIDE (HOE490) — Pharmaceutical form: 2 mg and 4 mg tablets Route of administration: oral
  Arms: glimepiride
Drug: SITAGLIPTIN — Pharmaceutical form: 100 mg tablets Route of administration: oral
  Arms: sitagliptin

SUMMARY:
Primary Objective:

To determine the superiority of glimepiride over sitagliptin in the reduction of HbA1c after 6 months of treatment in patients with monotherapy until the end of the trial.

Secondary Objective:

To evaluate the effect of glimepiride compared to sitagliptin in:

Glucose in fasting conditions; Postprandial glucose; Percentage of patients with HbA1c < 7% and < 6.5%; Symptomatic Hypoglycemia; Body weight; Percentage of withdrawal and percentage of patients with rescue therapy; Safety (adverse events and serious adverse events, hypoglycemia, vital signs and laboratory results).

ELIGIBILITY:
Inclusion criteria:

* Subject naïve to treatment
* HbA1c > 8.5 up to 11 %
* Lipid lowering therapy, antihypertensive, hormonal substitutes, thyroid hormone substitutes, and contraceptives are allowed as long as they are kept at a stable dosing

Exclusion criteria:

* Treatment with any oral antidiabetics or insulin
* Known type 1 Diabetes Mellitus
* Pregnant or breast feeding women
* Ketoacidosis history
* History of sensitivity to any of the active substances
* Renal dysfunction : serum creatinine > or = 1.5 mg/dL in male subjects > or = 1.4 mg/dL in female subjects
* Liver impairment (ALT, AST > 3-fold the upper limit of normal range)
* Systemic corticosteroid treatment 3 months prior to study or during the study
* Drug or alcohol abuse history
* Patients with history of acute coronary syndrome, cerebrovascular events/transient ischaemic attack in the last three months
* Presence of any condition (medical, psychological, social or geographic) current or previously seen that according to Investigators judgment jeopardizes the safety or restricts the participation of the patient during the study
* Neoplasias

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Actual)
Dates: Start 2009-07; Primary Completion 2010-10 (Actual); Study Completion 2010-10 (Actual)

PRIMARY OUTCOMES:
HbA1c | at baseline, week 12 and week 24
Fasting and postprandial glucose | at baseline, week 2, 4, 12 and 24

CONTACTS AND LOCATIONS:
Overall Officials: Judith Diaz, Study Director — Sanofi
Locations (2):
- Sanofi-Aventis Administrative Office, Guatemala City, Guatemala
- Sanofi-Aventis Administrative Office, Col. Coyoacan, Mexico